CLINICAL TRIAL: NCT04466735
Title: 6 Month Randomized Controlled Trial With D-beta-hydroxybutyrate in Mild Cognitive Impairment
Brief Title: BRain Energy Activation With Ketones to Prevent Alzheimer's Disease
Acronym: BREAK-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Alzheimer's Association (Other); Nestle Health Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-3448
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: MCI

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. First phase :Two parallel groups, one placebo, one active Second phase : All participants will be invited to take part in an open phase on the active product only.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators, participants and outcome assessors will be fully blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active group (Experimental): Participants will be on the active intervention for 6 months
  Interventions: Dietary Supplement: Active group
- Placebo Group (Placebo Comparator): Participants will be on the placebo intervention for 6 months
  Interventions: Dietary Supplement: Placebo group
- Open phase on active product (Active Comparator): At the end of the 6-month randomized controlled phase, participants will be unblinded and invited to continue on the active product for an additional 3 months.
  Interventions: Dietary Supplement: Active group

INTERVENTIONS:
Dietary Supplement: Active group — 2 x 12 g of EKS/day
  Arms: Active group; Open phase on active product
Dietary Supplement: Placebo group — Isocaloric placebo supplement with similar salt load but no EKS
  Arms: Placebo Group

SUMMARY:
A six month randomized controlled intervention with an exogenous ketone salt (EKS) supplement in mild cognitive impairment. Participants will receive 15 g of the supplement twice daily (equivalent to 24 g/day of EKS). Outcomes: brain energy metabolism, cognition, plasma biomarkers, brain imaging (volumetric, functional, structural) and quality of life will be analyzed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The participant must answer Yes to the question ''Do you think your memory is not as good as it was?''
* Have a MoCA Score between 20/30 and 26/30
* Have a QAF score of less than 9/30
* Understand, read and talk French
* Having good visual and hearing acuity

Exclusion Criteria:

* Major cognitive decline or neurodegenerative disease.
* Already consuming a daily medium chain triglyceride or ketone supplement.
* Soy, milk, gluten or allergy to the study product
* Controlled or uncontrolled diabetes
* Uncontrolled chronic disease
* Vitamin B12 deficit
* Clinical anomaly in the blood chemistry profile
* QSP-9 score over 19/27
* Taking an anti-cholinergic drugs
* Recent change in medication
* Active cancer in the last 2 years
* General anesthesia in the last 6 months
* history of alcohol abuse or dependence in the last 2 years
* Participation in other interventional or PET research project
* Unable to undergo an MRI or PET scan
* History of kidney stones or hypercalcemia
* History of cardiovascular events or insufficiency
* Renal failure and / or creatinine <58 umol or> 110 umol for men and <46 umol or> 92 umol for women or if the GFR (glomerular filtration rate) <60 ml / min / 1.73 m2
* Chronic disease of the digestive system or intestinal malabsorption (celiac disease, chronic pancreatitis, Crohn's disease, etc.)
* Body mass index <20 or voluntary weight loss of more than 5% in the last 6 months.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Acetoacetate brain uptake | 6 months
  CMRacac measured by PET Scan
Glucose brain uptake | 6 months
  CMRgluc measured by PET Scan

SECONDARY OUTCOMES:
Cognition | 0-3-6-9 months
Plasma biomarkers | 9 months
  glucose, fatty acids, ketones
Structural and functional brain measures | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rearsh Centre on Aging, Sherbrooke, Quebec, Canada